CLINICAL TRIAL: NCT05735860
Title: Die Nutzung Virtueller Realität Zur Behandlung Von Auftrittsangst
Brief Title: The Application of Virtual Reality Exposure Versus Relaxation Training in Music Performance Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 194/21-sc
Record Dates: First submitted 2022-12-14; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Music Performance Anxiety
MeSH Terms: interventions — Virtual Reality Exposure Therapy; Autogenic Training

STUDY DESIGN:
Intervention Model Description: randomized controlled / two-arm parallel assignment
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exposure Therapy (VRET) (Experimental)
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)
- Progressive Muscle Relaxation (PMR) (Active Comparator)
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy (VRET) — Four VRET sessions of approx. one hour each session taking place in an individual setting accompanied by a therapist. The participants wear a head-mounted display showing different musical performance scenarios (i.e. audition in a concert hall/ recording studio/ in front of a professional jury/ an audience/ a class of music students) that are selected individually by a previously standardized, graded exposure procedure.
  Arms: Virtual Reality Exposure Therapy (VRET)
Behavioral: Progressive Muscle Relaxation (PMR) — Four PMR sessions of approx. 45min each session taking place in an individual setting accompanied by a therapist. The sessions follow a previously standardized procedure.
  Arms: Progressive Muscle Relaxation (PMR)

SUMMARY:
The aim of the study is to investigate the effect of exposure treatment using virtual reality (VR) in musicians with performance anxiety compared to a relaxation technique on anxiety symptoms and corresponding cardiovascular parameters. The prospective, randomized clinical trial will include 46 musicians with musical performance anxiety (MPA). The experimental group will receive four exposure sessions in VR and the control group will receive four progressive muscle relaxation (PMR) sessions. Anxiety symptoms will be measured using a german version of the Performance Anxiety Questionnaire and a behavioral assessment test (BAT) before, after the treatment, and at 6-month follow-up. The cardiovascular reactivity will be assessed measuring the heart rate variability (HRV) throughout the BAT and the blood pressure before and after the BAT. Furthermore, blood and saliva samples will be collected before and after the BAT to assess endocrine stress parameters and epigenetic markers. The following hypotheses are derived: 1) Significant and lasting reduction of subjective MPA symptoms for the experimental group receiving VRET at T1 (post/ shortly after treatment) and T2 (follow-up/ 6 months after treatment) compared to T0 (pre/ before treatment). 2) Significant better reduction of subjective MPA symptoms for the experimental group receiving VRET compared to the control group receiving PMR at T1 (post/shortly after treatment) and T2 (follow-up/ 6 months after treatment) compared to T0 (pre/ before treatment). 3) The postulated effects in hypotheses 1 and 2 go along with a significantly higher HRV representing less cardiac stress during the BAT in case of a successful reduction of anxiety symptoms at T1 (post/ shortly after treatment) and T2 (follow-up/ 6 months after treatment) compared to T0 (pre/ before treatment).

ELIGIBILITY:
Inclusion Criteria:

* Music performance anxiety (MPA)

  * Reporting anxiety and/or avoidance of musical performance situations
  * Reporting psychological distress and/or impaired functioning due to the MPA
* Sufficient knowledge of the German language (to understand questionnaires and the therapy manual)
* Compliance with the covid-19-regulations for local study appointments
* Written informed consent

Exclusion Criteria:

* Substance use disorder
* Physiological contraindications for an exposure therapy (i.e. epilepsy, serious disorder of the cardiovascular system)
* Psychological contraindications for an exposure therapy (i.e. psychotic disorder, substance dependence, borderline personality disorder, acute suicidality)
* Use of sedative medication or tranquilizers (i.e. beta-blockers) for the therapy appointments
* Claustrophobia
* Blood-injection-injury type phobia
* Instrument not portable, too big or not playable while standing (i.e. piano, drums, harp, double bass)
* Not able to play the instrument blindfold
* Current psychotherapy because of the MPA
* Recent (< 6 months ago) psychotherapy because of the MPA

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
German Version of the Performance Anxiety Questionnaire (Fehm, 2002) | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring subjective MPA symptoms for solo and ensemble performances by assessing the total score for the scale solo performance (0-80) and the total score for the scale ensemble performance (0-80). Higher scores indicate more symptoms of music performance anxiety.
Heart rate variability | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring the cardiac reactivity throughout the BAT in virtual reality

SECONDARY OUTCOMES:
Subjective Units of Distress (SUDs) during the BAT | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring subjective MPA (0-100) in the BAT in virtual reality. Higher scores indicate a higher level of anxiety.
Social Interaction Anxiety Scale (SIAS) | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring symptoms of social anxiety or distress specifically when talking or meeting others. A higher total score (0-80) indicates more symptoms of social anxiety.
Social Phobia Scale (SPS) | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring symptoms of social phobia specifically in anticipation of or when actually being observed by others and when engaging in activities in the presence of others. A higher total score (0-80) indicates more symptoms of social anxiety.
Beck Depression Inventory (BDI-II) | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring symptoms of depression. A higher total score (0-63) indicates more symptoms of depression.
Beck Anxiety Inventory (BAI) | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring symptoms of anxiety. A higher total score (0-63) indicates more symptoms of anxiety.
Anxiety Sensitivity Index (ASI-3) | Only one assessment at T0 (pre/ before treatment)
  Measuring anxiety sensitivity. A higher total score (0-56) indicates a higher level of anxiety sensitivity.
State Trait Anxiety Inventory - Trait (STAI-Trait) | Only one assessment at T0 (pre/ before treatment)
  Measuring trait anxiety. A higher total score (20-80) indicates a higher level of trait anxiety.
Childhood Trauma Questionnaire (CTQ) | Only one assessment at T0 (pre/ before treatment)
  Measuring childhood-history of abuse and neglect by assessing the total scores for the scales Emotional Neglect (7-35), Sexual Abuse (5-25), Physical Abuse and Neglect (7-35), and Emotional Abuse (5-25). Higher Scores indicate a higher level of childhood abuse and/or neglect.
Immersive Tendencies Questionnaire (ITQ) | Only one assessment at T0 (pre/ before treatment)
  Measuring immersive tendencies. Higher scores on the scales Focus (5-35), Implication (5-25), Emotion (4-28), Joy (3-31) and a higher total score (17-119) indicate a higher level of immersive tendencies.
Uncertainty Tolerance Scale (UGTS) | Only one assessment at T0 (pre/ before treatment)
  Measuring uncertainty tolerance. A higher total score (8-48) indicates a higher level of uncertainty tolerance.
Positive and Negative Affect Schedule (PANAS) | Change from before to after (approx. 45min later) the BAT in VR at T0 (pre/ before treatment), T1 (post/ approx. one week after treatment) and T2 (follow-up/ 6 months after treatment)
  Measuring state affect. Higher scores on the scales Positive Affect (10-50) and Negative Affect (10-50) indicate a higher level of positive or negative state affect.
Blood pressure | Change from before to after (approx. 30min later) the BAT in VR at T0, T1 and T2; and changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring cardiac stress
Heart rate | Change from before to after (approx. 30min later) the BAT in VR at T0, T1 and T2; and changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring cardiac stress
Salivary cortisol hormone | Change from before to after (approx. 30min later) the BAT in VR at T0, T1 and T2; and changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring the psychophysiological stress response
Neuropeptides | Changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Analysis of neuropeptides with modulating effects on humoral and behavioral stress response, and myocardial as well as autonomic nerve system function, such as Atrial natriuretic Polypeptide (ANP), neuropeptide Y (NPY), Oxytocin (OCT), salivary Alpha-Amylase (sAA).
Epigenetic Targets | Change from before to after (approx. 30min later) the BAT in VR at T0, T1 and T2; and changes from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  mDNA analysis of the candidate genes related to the endocrine stress reactivity (NR3C1, FKBP5, CRHR1) and DNAm analysis of Norepinephrine Transporter (NET) and Oxytocin Receptor (OXTR) genes due to their implication in the regulation of autonomous function and social anxiety
Kenny Music Performance Anxiety Inventory-Revised (K-MPAI-R) | Change from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring performance anxiety in musicians. A higher total score (0-240) indicates a higher level of music performance anxiety.
Questionnaire on safety- and avoidance behaviors for musicians (Mumm et al., 2020) | Change from T0 (pre/ before treatment) to T1 (post/ approx. one week after treatment) and from T0 (pre/ before treatment) to T2 (follow-up/ 6 months after treatment)
  Measuring the use of safety and avoidance behaviors in musicians. A higher total score (0-215) indicates a higher use of safety- and avoidance behaviors to reduce anxiety in performance situations.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Psychosomatics, and Psychotherapy, Center for Mental Health, University Hospital of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Derived] Bellinger D, Wehrmann K, Rohde A, Schuppert M, Stork S, Flohr-Jost M, Gall D, Pauli P, Deckert J, Herrmann MJ, Erhardt-Lehmann A. The application of virtual reality exposure versus relaxation training in music performance anxiety: a randomized controlled study. BMC Psychiatry. 2023 Aug 1;23(1):555. doi: 10.1186/s12888-023-05040-z. PMID 37528410